CLINICAL TRIAL: NCT00543452
Title: Effect of Oxygen on Core Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swedish Heart Lung Foundation (Other)
Responsible Party: Karl Franklin, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 03-567
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-03

CONDITIONS: Cardiac Disease; Cheyne-Stokes Respiration
MeSH Terms: conditions — Heart Diseases; Cheyne-Stokes Respiration | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- oxygen (Active Comparator): 4 liters of oxygen a minute
  Interventions: Other: Oxygen
- air (Placebo Comparator): 4 liters of room air
  Interventions: Other: Air from a placebo oxygen delivery

INTERVENTIONS:
Other: Oxygen — 4 liters of oxygen a minute
  Arms: oxygen
Other: Air from a placebo oxygen delivery — 4 liters a minute of air from a placebo device
  Arms: air

SUMMARY:
Study of the effect of oxygen on the frequency of central apnea, sleep and body temperature in patients with a cardiac disease

ELIGIBILITY:
Inclusion Criteria:

* Cardiac disease and Cheyne-Stokes respiration and controls without Cheyne-Stokes respiration

Exclusion Criteria:

* Obstructive sleep apnea

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Core temperature | One day
  This is an experitmetal study. Subjects receive oxygen or placebo-air during one night in random order. Outcome measure, i.e.core temperatue is measured continuously during this night with ongoing treatment of oxygen or placebo-air

SECONDARY OUTCOMES:
Sleep stages, apnea-hypopnea index | One day
  This is an experitmetal study. Subjects receive oxygen or placebo-air during one night in random order. Outcome measure, i.e.the amount of differernt sleep stages, total sleep time and apnea-hypopnea index is measured during this night with ongoing treatment of oxygen or placebo-air

CONTACTS AND LOCATIONS:
Overall Officials: Karl A Franklin, MD, PhD, Principal Investigator — Dept Respiratory Medicine, University Hospital, Umeå
Locations (1):
- Dept of respiratory medicine, Umeå, Sweden